CLINICAL TRIAL: NCT01157546
Title: Continuous Transversus Abdominis Plane (TAP) Block for Open Radical Prostatectomy. A Double Blind Randomized Study.
Brief Title: TAP Block for Open Radical Prostatectomy.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low recruitment rate. In our center, open radical prostatectomies have been almost completely replaced by robotic prostatectomies.
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Gabriele Baldini, MD, MSc, Assistant Professor, MD, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GEN-10-012
Record Dates: First submitted 2010-06-30; First posted 2010-07-07 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Opioid Consumption; Incidence of Nausea and Vomiting; Postoperative Pain; Assessment of Recovery
MeSH Terms: conditions — Vomiting; Pain, Postoperative | interventions — Saline Solution; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): group A (control) will receive a bolus of normal saline (20 mL per side) followed by a continuous infusion of normal saline (7 ml/h per side) via both TAP catheters.The infusions will be started after the bolus doses and continued postoperatively for 48 hours.
  Interventions: Procedure: Normal saline via TAP catheters
- TAP (Experimental): group B (TAP) will receive a bolus of lidocaine 1% with epinephrine 1:200 000 (20 mL per side) followed by a continuous infusion of ropivacaine 0.2% (7 mL/h per side) via TAP catheters. The infusions will be started after the bolus doses and continued postoperatively for 48 hours.
  Interventions: Procedure: Lidocaine via TAP catheters

INTERVENTIONS:
Procedure: Normal saline via TAP catheters — A bolus of normal saline (20 mL per side) followed by a continuous infusion of normal saline (7 ml/h per side. The infusions will be started after the bolus doses and continued postoperatively for 48 hours.
  Other Names: 0.9% normal saline; NSS
  Arms: Control
Procedure: Lidocaine via TAP catheters — A bolus of lidocaine 1% with epinephrine 1:200 000 (20 mL per side) followed by a continuous infusion of ropivacaine 0.2% (7 mL/h per side). The infusions will be started after the bolus doses and continued postoperatively for 48 hours.
  Other Names: Xylocaine
  Arms: TAP

SUMMARY:
This is a prospective, double blind, randomized study is proposed in patients undergoing open radical prostatectomy: its objective is to establish whether continuous bilateral TAP blocks would provide adequate perioperative analgesia, decrease opioid consumption, reduce the incidence of opioid-related side effects, and facilitate surgical recovery (in terms of PACU and hospital discharge).

DETAILED DESCRIPTION:
Open prostatectomy is a surgical procedure performed by urologists to excise the prostate. This is achieved by a 10-cm vertical incision starting below the umbilicus and reaching the pubic area. Patients are hospitalized for 3-4 days: one of the criteria for safe discharge includes Visual Analogue Scale (VAS) for pain below 3 at rest. For postoperative pain control, patients receive patient-controlled opioid analgesia (PCA) with morphine. The average amount of morphine used in the first 24 h varies between 30 and 50 mg. Although this technique is widely used, side effects (sedation, ileus, pruritus) are commonly encountered with opioid administration. Thus alternative analgesic techniques such as epidural analgesia and wound infiltration have been used with some success. However adverse events have also been reported with these techniques (lower limb motor block with epidural; infection wound infiltration).

In the last 10 years, a new technique, the transversus abdominis plane (TAP) block, which anesthetizes the thoracolumbar nerves (intercostal, subcostal and first lumbar nerves), has been described. The thoracolumbar nerves provide sensory innervation to the anterolateral abdominal wall. The traditional technique for TAP blocks is performed with a blunt needle in the Triangle of Petit. The latter is delineated caudally by the iliac crest, posteriorly by the latissimus muscle and anteriorly by the external oblique. Two distinct pops can be felt as the needle crosses the fascial extensions of the external oblique and the internal oblique muscle, respectively. Thus the second pop usually signifies that the needle tip has reached the TAP. Although the traditional technique has been used to provide postoperatively analgesia for bowel surgery, hysterectomy and Cesarian Section, the position of the Triangle of Petit varies greatly thus making it difficult to palpate in obese patients. In 2007, there was a study describing an ultrasound-guided technique for TAP blocks: these authors advocated using ultrasonography to locate the TAP along the mid-axillary line above the iliac crest. This ultrasound-guided technique has been subsequently used to provide postoperative analgesia for laparoscopic cholecystectomy, appendicectomy and Cesarian Section. This technique has been shown to spare opioids in the postoperative period therefore facilitating an accelerated discharge and superior pain relief.

In our institution, the TAP block, either as a single shot or as a continuous catheter infusion, is used for abdominal and urological surgery when epidural blockade is not feasible.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and over
* ASA class 1, 2
* Elective open radical prostatectomy

Exclusion Criteria:

* Any history or signs of cardiac, hepatic and renal failure. Patients with raised serum LFTs and serum creatinine outside normal range
* Any chronic use of opioid analgesic
* Morbid obesity (BMI>40)
* History of allergic reactions to any of the study medications and the medications used for the trial
* Pregnancy
* Previous abdominal surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Postoperative morphine consumption | at 24 hour after surgery

SECONDARY OUTCOMES:
Incidence of nausea and vomiting | at 2, 12, 24 and 48 hour after surgery
VRS for pain at rest, during ambulation and coughing | at 2, 12, 24 and 48 hour after surgery
Assessment of recovery | at 24 hours after the surgery and every 24 hours until patients are discharged.
  Assessment of recovery (two-minute walking test, Miles scale) and time out of bed (sitting or walking will be measured every day until hospital discharge.
Postoperative morphine consumption | at 2, 12 and 48 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Franco Carli, Professor, Principal Investigator — McGill University Healt Centre, Department of Anesthesia
Locations (1):
- McGill University Health Centre, Montreal General Hospital, Montreal, Quebec, Canada